CLINICAL TRIAL: NCT00407394
Title: Randomized Double Blind Placebo Controlled Trial of Amoxycillin in the Treatment of Non-Severe Pneumonia With Wheeze in Children Aged 2- 59 Months of Age: A Multi-Centric Study
Brief Title: Indiaclen Short Course Amoxycillin Therapy for Pneumonia With Wheeze
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King George's Medical University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9998
Record Dates: First submitted 2006-12-02; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Non-Severe Pneumonia With Wheeze
Keywords: Pneumonia; Wheezing; Treatment; Children; India
MeSH Terms: conditions — Pneumonia; Respiratory Sounds | interventions — Amoxicillin

INTERVENTIONS:
Drug: Amoxycillin

SUMMARY:
Background: The current Integrated management of childhood infections (IMCI) algorithm prescribes that children with wheeze and fast breathing presenting to first level health facilities are given antibiotics if they continue to have fast breathing after two doses of bronchodilator. The primary purpose of the algorithm is to prevent mortality due to bacterial pneumonia. However, an unknown proportion of children managed in this fashion will have a viral related wheezing illness or asthma rather than pneumonia. Although it is unlikely that wheezing syndromes are a significant cause of mortality for children in developing countries, these algorithms are likely to result in unnecessary administration of antibiotics as well as inadequate treatment of recurrent wheezing illness. We do not have clear evidence about whether antibiotics can be withheld in some categories of children with wheeze. It is clear that wheeze can occur in bacterial infection and in addition co-infection with virus and bacteria has been well demonstrated in several studies of pneumonia etiology in children. Although some studies have found that children with more severe disease or who are blood culture positive are more likely to be febrile at presentation, this sign is not sufficiently sensitive or specific to determine whether antibiotics should be administeredSetting: The study will be conducted in eight medical colleges situated in Lucknow, Nagpur, New Delhi, Mumbai, Chennai, Trivandrum, Vellore, and Chandigarh. Design: This will be a multicentric, randomized, double blind efficacy trial. . Hypothesis: The primary hypothesis is that the use of oral amoxycillin for three days would be as effective, in terms of clinical cure on day 4 as compared to use of oral placeboMain objective: To compare the proportion of children aged 2 to 59 months presenting with non-severe pneumonia with wheeze whose respiratory rate does not fall below the age specific cut-off after three doses of nebulized salbutamol, that achieve clinical cure on day 4 on 3 day of treatment with oral amoxycillin versus placebo.Inclusion criteria: Children aged 2-59 months with non-severe pneumonia based on WHO criteria of respiratory rate above the age specific cut-off, audible / ausculatory wheeze. Exclusion criteria: Children with severe disease, received any documented antibiotic treatment in the past 48 hours, diagnosed asthmatic on maintenance therapy, complicating acute non-pulmonary or chronic illness, known drug allergy, hospitalization in the past 2 weeks, history of measles within the last month, known immunodeficiency disorder, prior enrollment in the study, residing in areas not accessible for follow-up or whose guardian refuses to consent for the study. Sample size: Has been calculated to test the null hypothesis. There will be 950 children in each arm. Thus each site is required to recruit a minimum of 225 cases over 18 months.

DETAILED DESCRIPTION:
Background: The World Health Organizations acute lower respiratory infections (ALRI) management algorithms depend primarily on two key clinical signs: elevated respiratory rate and chest indrawing. The current Integrated management of childhood infections (IMCI) algorithm prescribes that children with wheeze and fast breathing presenting to first level health facilities are given antibiotics if they continue to have fast breathing after two doses of bronchodilator. The primary purpose of the algorithm is to prevent mortality due to bacterial pneumonia. However, an unknown proportion of children managed in this fashion will have a viral related wheezing illness or asthma rather than pneumonia. Although it is unlikely that wheezing syndromes are a significant cause of mortality for children in developing countries, these algorithms are likely to result in unnecessary administration of antibiotics as well as inadequate treatment of recurrent wheezing illness. In both developed and developing countries respiratory syncytial virus is the predominant etiological agent responsible for bronchiolitis and wheezing illness in the first two years of life. Moreover data from several studies demonstrates that respiratory syncitial virus (RSV) infection and the bronchiolitis syndrome are a major component of the total ALRI in children living in developing countries. The relevant literature on therapy includes studies in which children were labelled as bronchiolitis and others in which children were classified as wheezing illness.We do not have clear evidence about whether antibiotics can be withheld in some categories of children with wheeze. It is clear that wheeze can occur in bacterial infection and in addition co-infection with virus and bacteria has been well demonstrated in several studies of pneumonia etiology in children. Although some studies have found that children with more severe disease or who are blood culture positive are more likely to be febrile at presentation, this sign is not sufficiently sensitive or specific to determine whether antibiotics should be administered.There has been extensive debate about whether infants and young children in the first year of life respond to bronchodilator therapy. Proposed reasons for a lack of response have included: immaturity of bronchiolar smooth muscle, increased dynamic airway closure and relatively larger degrees of mucosal edema. A literature search between 1980 and 2000 reveals five randomized placebo controlled trials of beta agonist administered to acutely wheezing infants in which clinical outcomes were determined. Overall these studies support the hypothesis that children aged less than 12 to 18 months are less responsive to bronchodilator therapy than older children. However, they also demonstrate that use of inhaled short acting bronchodilators for the acute treatment of wheeze offers some benefits for clinical outcomes even in this young age group. The benefits of beta agonists may be restricted to children with recurrent wheezing and at most provide a very small clinical benefitSetting: The study will be conducted in eight medical colleges situated in New Delhi, Chandigarh, Lucknow, Mumbai, Nagpur, Chennai, Vellore and Trivandrum. Design: This will be a multicentric, randomized, double blind efficacy trial. Block randomization will be done in Dept. of Pharmacology, KGMU, Lucknow, which is not the coordinating center for the trial. Blocks will be generated in mixed batches. The medicines will be then placed in by the pharmacy according to the intervention type determined by the pharmacy. Two hundred and twenty five random numbers will be generated in blocks of varying lengths for each of the nine sites.OutcomesPrimary: Clinical Cure: Respiratory rate below agerate below ages specific cut-off (<50 bpm in infants <1 year and <40 bpm in ages 12 - 59 months) and absence of auscultatory as well as audible wheeze.Secondary: Response to nebulization: Respiratory rate below age specific cut-off (<50 bpm in infants <1 year and <40 bpm in ages 12 - 59 months) after a maximum of three doses of nebuliaztion with salbutamol, auscultaroy wheeze may or may not be present. But there is no audible wheeze.Clinical failure of therapy: Any signs of severe pneumonia or severe disease; chest in drawing, convulsions, drowsiness or inability to drink at any time; Respiratory rate above age specific cut-off on day 4 or after that (with or without wheeze);Oxygen saturation on pulse oximetry <90% on day 4 or after that; Documented axillary temperature > 101 degrees Fahrenheit. In addition, children who die within the follow-up period of 14 days or are lost to follow-up on day 4 will also be considered as failed.Clinical relapse at day 7- 15: Signs of severe pneumonia or very severe disease among cases who were clinically cured on day 4 follow-up.Hypothesis: The primary hypothesis is that the use of oral amoxycillin for three days would be as effective, in terms of clinical cure on day 4 as compared to use of oral placebo. Intervention: Amoxycillin tablets (125 mg) or placebo They will be used after dissolving in 5 ml of clean water. The medicines will be given according to the weight of the child as follows:q 4 - 6 KG ½ tablet thrice a dayq 7 - 10 KG 1 tablet thrice a dayq 11 - 15 KG 1 ½ tablet thrice a dayq 16 - 20 KG 2 tablets thrice a dayMain objective: To compare the proportion of children aged 2 to 59 months presenting with non-severe pneumonia with wheeze whose respiratory rate does not fall below the age specific cut-off after three doses of nebulized salbutamol, that achieve clinical cure on day 4 on 3 day of treatment with oral amoxycillin versus placeboSecondary objectives: Among all cases of non-severe pneumonia with wheeze1. To assess the proportion of children aged 2 to 59 months presenting with non-severe pneumonia with wheezing audible wheeze2. To assess the proportion of children aged 2 to 59 months presenting with non-severe pneumonia with wheezing who respond to up to three doses of nebulization with salbutamol.Among cases of non-severe pneumonia with wheeze aged 2 to 59 months who respond to three doses of salbutamol3. To assess the proportion of who fail therapy at day 4 of the initial successful bronchodilator therapy with inhaled salbutamol.4. To assess the proportion relapse at day 11- 14 of the initial successful bronchodilator therapy with inhaled salbutamol.5.To compare the cost of treatment of clinical failures and relapses among those treated with oral salbutamol.6 .To assess the association of bronchodilator response with age, season, number of previous wheezing episodes, audible versus auscultatory wheeze and family history of asthma.7.To assess the association of relapse in children who showed improvement after being treated with inhaled salbutamol, with age, respiratory syncytial virus (RSV) isolation, season, number of previous wheezing episodes, audible versus auscultatory wheeze and family history of asthma.Among cases of non-severe pneumonia with wheeze aged 2 to 59 months who do not respond to three doses of salbutamol8.To compare the proportion of children who are judged to be clinically cured after 3 days of treatment but who relapse within the next 11-14 days observation on 3-day treatment with oral amoxycillin versus placebo.9.To compare the cost of treatment of clinical failures and relapses among those treated with oral amoxycillin or placebo.10. To assess the association of clinical failure on day 4 with age, respiratory syncytial virus (RSV) isolation, season, number of previous wheezing episodes, audible versus auscultatory wheeze, family history of asthma and randomization to amoxycillin therapy.Inclusion criteria: Children aged 2-59 months with non-severe pneumonia based on WHO criteria of respiratory rate above the age specific cut-off, audible / ausculatory wheeze, accessible to follow up, whose guardians give written informed consent.Exclusion criteria: Children with severe disease, received any documented antibiotic treatment in the past 48 hours, diagnosed asthmatic on maintenance therapy, complicating acute non-pulmonary or chronic illness, known drug allergy, hospitalization in the past 2 weeks, measles or history of measles within the last month, known immunodeficiency disorder, prior enrollment in the study, residing in areas not accessible for follow-up or whose guardian refuses to consent for the study. Radiological Pneumonia on X-Ray.Sample size: Two modes of therapies will be assumed to be equal if the failure rate in new regimen is not more than 17%. So each site will be required to recruit and follow up 225 cases in each arm over 18 months. Thus there will be 950 children in each arm.Policy relevance: The present study plans to evaluate the role of antibiotic in children with non-severe pneumonia presenting with wheeze. It will define the patient and disease characteristics associated with clinical failure and the need for antibiotics. The results of the study will formulate policy to use antibiotics in children with non-severe pneumonia and wheeze.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-59 months with non-severe pneumonia based on WHO criteria of respiratory rate above the age specific cut-off, audible / ausculatory wheeze, accessible to follow up, whose guardians give written informed consent.

Exclusion Criteria:

* Children with severe disease, received any documented antibiotic treatment in the past 48 hours, diagnosed asthmatic on maintenance therapy, complicating acute non-pulmonary or chronic illness, known drug allergy, hospitalization in the past 2 weeks, measles or history of measles within the last month, known immunodeficiency disorder, prior enrollment in the study, residing in areas not accessible for follow-up or whose guardian refuses to consent for the study. Radiological Pneumonia on X-Ray.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000
Dates: Start 2004-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Clinical Cure: Respiratory rate below age specific cut-off (<50 bpm in infants <12 months and <40 bpm in 12 - 59 months of age).

SECONDARY OUTCOMES:
Clinical failure: Any signs of severe pneumonia or severe disease; chest in drawing, convulsions, drowsiness or inability to drink at any time; Respiratory rate above age specific cut-off on day 4 or after that; Oxygen saturation on pulse oximetry <90%

CONTACTS AND LOCATIONS:
Overall Officials: Shally Awasthi, MD, Principal Investigator — King George's Medical University, Lucknow, India
Locations (1):
- King George's Medical University, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Awasthi S, Agarwal G, Kabra SK, Singhi S, Kulkarni M, More V, Niswade A, Pillai RM, Luke R, Srivastava NM, Suresh S, Verghese VP, Raghupathy P, Lodha R, Walter SD. Does 3-day course of oral amoxycillin benefit children of non-severe pneumonia with wheeze: a multicentric randomised controlled trial. PLoS One. 2008 Apr 23;3(4):e1991. doi: 10.1371/journal.pone.0001991. PMID 18431478